CLINICAL TRIAL: NCT07401966
Title: Amputations in Childhood and Neuropathic Pain
Acronym: NAPE
Status: Not yet recruiting | Type: Observational
Sponsor: Hopitaux de Saint-Maurice (Other)
Responsible Party: Sponsor
Other Study IDs: NAPE; 2025-A02122-47 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2026-02-03; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pediatric; Neuropathic Pain; Phantom Limb Pain; Amputation
MeSH Terms: conditions — Neuralgia; Phantom Limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric limb amputation cohort: This cohort includes children and adolescents aged 5 to 18 years who underwent limb amputation during childhood and are followed at a specialized pediatric limb anomaly referral center.
  Participants are evaluated at a single time point using retrospective medical record data and standardized questionnaires administered during routine follow-up visits, without any modification of standard clinical care.

SUMMARY:
This observational study aims to assess the presence of neuropathic pain in children and adolescents who underwent limb amputation during childhood.

The study focuses on two types of neuropathic pain: phantom limb pain and residual limb pain. It also evaluates quality of life and functional autonomy in this population and explores potential associations between neuropathic pain, autonomy, quality of life, and age at amputation.

Using a mixed retrospective and prospective design, data are collected from medical records and standardized questionnaires administered during routine follow-up visits at a specialized pediatric limb anomaly center. The study seeks to improve understanding of neuropathic pain after pediatric amputation and its impact on daily functioning.

DETAILED DESCRIPTION:
Pediatric limb amputations are rare and may occur in the context of trauma, infection, tumors, or congenital malformations. In some congenital conditions, such as proximal femoral focal deficiency, therapeutic amputation may be proposed to improve prosthetic fitting, functional outcomes, and autonomy. One of the potential complications associated with limb amputation is the development of neuropathic pain, including phantom limb pain and residual limb pain. While these conditions are well documented in adults, their prevalence and impact in pediatric populations remain poorly understood.

Neuropathic pain may interfere with prosthetic use, functional abilities, quality of life, and long-term autonomy. In children who undergo amputation for functional purposes, the presence and consequences of neuropathic pain are important factors to consider when weighing the expected benefits of surgery. Early identification and management of neuropathic pain may also allow better anticipation and implementation of preventive or therapeutic strategies.

This monocentric observational study aims to describe the presence of neuropathic pain in children and adolescents who underwent limb amputation during childhood. Neuropathic pain is assessed using validated questionnaires, distinguishing between phantom limb pain and residual limb pain. The study also evaluates quality of life and functional autonomy using age-appropriate standardized assessment tools.

In addition, the study explores associations between neuropathic pain and functional autonomy, quality of life, age at amputation, and preoperative preventive treatments when applicable. Data are collected through a mixed retrospective and prospective approach, combining extraction of medical record information and a single administration of questionnaires during routine follow-up visits. No intervention or modification of standard clinical care is performed.

By providing descriptive data on neuropathic pain and its functional consequences after pediatric amputation, this study aims to contribute to improved clinical decision-making, pain management strategies, and long-term follow-up of children with limb amputations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 5 and 18 years (inclusive) (Piaget's concrete operational stage to be able to complete the self-assessment questionnaires)
* Patients who underwent amputation before the age of 15 for girls and 16 for boys (average age of completion of lower limb growth)
* Patients who have not undergone surgery on the amputated limb for at least one year (to avoid bias, as any surgery involving incision can cause temporary neuropathic pain unrelated to the amputation)
* Have obtained the signature of the non-objection form by both parents/legal guardians
* Have obtained the child's consent (verbal consent but recorded)
* Be affiliated with a health insurance plan.

Exclusion Criteria:

* Patients who do not speak French
* Patients whose cognitive abilities are insufficient (as determined by a clinician or reported by parents) to be able to complete self-assessment questionnaires
* Patients undergoing chemotherapy (due to transient neuropathic pain)
* Patients who have received chemotherapy and whose side effects have not yet subsided (on a case-by-case basis depending on the chemotherapy used)
* Patients who have received chemotherapy causing neuropathic pain due to this treatment that has not disappeared.
* Patients placed under protective custody.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of children and adolescents aged 5 to 18 years who underwent limb amputation during childhood and are followed at a specialized pediatric referral center for limb anomalies.
  Participants include individuals with upper limb and/or lower limb amputation, regardless of the etiology of amputation. The study population includes both prosthesis users and non-prosthesis users. Data are collected using retrospective medical record review and a single prospective assessment with standardized questionnaires administered during routine follow-up visits, without any modification of standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-11-09 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Presence of neuropathic pain after pediatric limb amputation | Single assessment at study inclusion (variable time after amputation)
  Presence of neuropathic pain assessed using the DN4 questionnaire, including phantom limb pain and residual limb pain. A DN4 score of 4 or higher is considered indicative of neuropathic pain.

SECONDARY OUTCOMES:
Type of neuropathic pain after pediatric limb amputation | At study inclusion
  Type of neuropathic pain reported after limb amputation, distinguishing phantom limb pain and residual limb pain, assessed using the DN4 questionnaire.
Health-related quality of life | At study inclusion
  Health-related quality of life assessed using the SF-15 Generic Core Scales questionnaire, adapted to the participant's age, in children and adolescents with limb amputation.
Locomotor capability in lower limb amputees | At study inclusion
  Locomotor capability assessed using the Locomotor Capability Index (LCI) in children and adolescents with lower limb amputation. The LCI score is analyzed in prosthesis users, for whom the scale is validated. For non-prosthesis users, a descriptive analysis of individual items is performed.
Upper limb functional ability | At study inclusion
  Upper limb functional ability assessed using the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire in children and adolescents with upper limb amputation.
Association between neuropathic pain and quality of life | At study inclusion
  Association between the presence of neuropathic pain and health-related quality of life after pediatric limb amputation.
Association between neuropathic pain and functional outcomes | At study inclusion
  Association between the presence of neuropathic pain and functional outcomes, including locomotor capability in lower limb amputees and upper limb functional ability in upper limb amputees.
Association between neuropathic pain and age at amputation | At study inclusion
  Association between the presence of neuropathic pain and age at the time of limb amputation.

CONTACTS AND LOCATIONS:
Overall Officials: Margaux MM Modjbafan, Principal Investigator — Hôpitaux Paris Est Val-de-Marne, centre de référence des malformations des membres, Saint-Maurice 94410; Maïwenn MF Feldmann, Study Director — Hôpitaux Paris Est Val-de-Marne, centre de référence des malformations des membres, Saint-Maurice 94410
Locations (1):
- Hôpitaux Paris Est Val-de-Marne - Centre de Référence des Malformations des Membres, Saint-Maurice, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the observational design of the study, the pediatric population involved, and the need to protect sensitive medical and functional data. Data are pseudonymized and handled in accordance with applicable data protection regulations, and no public data-sharing plan is planned.